CLINICAL TRIAL: NCT02267473
Title: A Multicenter, Prospective, Observational Study of Patients With Chronic Hepatitis B Under Various Oral Nucleos(t)Ide Treatment With Intermittent Assessment of Kidney Function
Brief Title: Hepatitis B Patients Under Oral Nucleos(t)Ide Treatment With Intermittent Assessment of Kidney Function
Acronym: BONIKA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Vermehren, MD, Johann Wolfgang Goethe University Hospital
Other Study IDs: JWGUHMED1-008
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — spontaneous urine sample to test for proximal tubular function
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with chronic Hepatitis B who are under oral antiviral treatment for at least 6 months at study start will be monitored once yearly for kidney function changes within their routine outpatient visit. Therefore urine samples will be collected and some additional blood test will be done within the routine blood sampling.

DETAILED DESCRIPTION:
This non-interventional, long-term observational cohort study will evaluate demographic, clinical, biochemical and virological parameters of outpatients with chronic Hepatitis B who are under oral antiviral treatment with an approved Nucleos(t)ide for > 6 months at study inclusion.

During their routine outpatient visits annually an assessment of their kidney function especially for a proximal tubular dysfunction will be performed and their comedication will be explored. Patients included in the study are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* chronic Hepatitis B Virus infection
* indication for an antiviral treatment due to the recent german Hepatitis B guidelines and oral intake of an approved Nucleos(t)ide for a minimum of 6 months at inclusion
* ALT < 2 x UNL (upper normal limit) at study inclusion
* age 18 - 89 years
* signed informed consent form

Exclusion Criteria:

* coinfection with Hepatitis D Virus (HDV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV)
* Comorbidities that will hinder the study performance (e.g. malignancies, relevant psychiatric disorder)
* hepatocellular carcinoma or hepatic metastases
* legally incapacitated patients

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic Hepatitis B under oral antiviral treatment with an approved Nucleos(t)ice for a minimal duration of 6 months at study inclusion
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Kidney Function | 5 Years
  Reproducible change in creatinine >0.3mg/dl or signs of proximal tubular dysfunction

SECONDARY OUTCOMES:
Kidney relevant Comorbidities | 5 Years
  Proportion of patients with kidney relevant comorbidities like arterial hypertension, diabetes mellitus, gout
Kidney relevant Comedication | 5 Years
  Relevance of Comedication e.g. Non Steroidal AntiInflammatory Drugs (NSAIDs) to the kidney function under oral antiviral treatment of chronic Hepatitis B
HBV-DNS | 5 Years
quantitative HBs Antigen | 5 Years
Mitochondrial Toxicity | 5 Years
  Signs of mitochondrial toxicity under oral antiviral Hepatitis B Treatment like Lipodystrophy or changed fat metabolism

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Klinikum der J. W. Goethe-Universität, Frankfurt